CLINICAL TRIAL: NCT01317667
Title: Phase 1 Escalating, Multiple-Dose Study to Evaluate the Safety and Immunogenicity of Recombinant Ricin Toxin A-Chain 1-33/44-198 (rRTA 1-33/44-198) Vaccine (RVEc™) in Healthy Adults
Brief Title: Safety and Immunogenicity Study of Recombinant Ricin Toxin A-Chain Vaccine (RVEc™)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S-10-0002, FY09-03, A-16390
Record Dates: First submitted 2011-03-09; First posted 2011-03-17 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Ricin
Keywords: Ricin; RVEc
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): RVEc vaccine 20 μg/dose x 3 doses
  Interventions: Biological: RVEc
- Group 2 (Experimental): RVEc vaccine 50 μg/dose x 3 doses
  Interventions: Biological: RVEc
- Group 3 (Experimental): RVEc vaccine 100 μg/dose x 1 dose
  Interventions: Biological: RVEc

INTERVENTIONS:
Biological: RVEc
  Other Names: Recombinant Ricin Toxin A-Chain 1-33/44-198 (rRTA 1-33/44-198) Vaccine

SUMMARY:
This study is a Phase 1, escalating, multiple-dose, single-center study to evaluate the safety and immunogenicity of the RVEc vaccine.

The two principal hypotheses to be tested are: RVEc vaccine will display an acceptable safety profile as determined by adverse event data and RVEc vaccine will elicit ELISA immunoglobulin G (IgG) titers greater than or equal to 1:500 and toxin-neutralizing antibody (TNA) anti-ricin toxin-neutralizing antibody titers greater than or equal to 1:50 in vaccine recipients.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be 18-50 years old.
* Subjects must weigh at least 110 pounds.
* Subjects must be in good health as judged from medical history, physical examination, EKG and chest x-ray, complete blood count (CBC) with differential, clinical chemistries, urinalysis, hepatitis serology, and HIV antibody test, and be medically cleared for participation by an investigator. If any HIV or hepatitis testing is positive, the individual will be provided with counseling and referral for health care.
* Females of childbearing potential must have a negative pregnancy test on vaccination day before each dose and agree to not become pregnant or breastfeed for 3 months after the last dose of the vaccine and be willing to use a reliable form of contraception during the study.
* Study subjects must read and sign an approved informed consent.
* Study subjects must be willing to complete a subject diary card after each vaccination.
* Study subjects must be willing to return for all follow-up visits.
* Study subjects must agree to report any adverse event (AE) that may or may not be associated with administration of the investigational product through the 9-month follow-up visit. Study subjects will report all serious adverse events for the duration of the study.

Exclusion Criteria:

* Body weight less than 110 pounds.
* Acute or chronic medical conditions or immunodeficiency from a medical condition or medical treatment, medications, or dietary supplements that, in the investigator's opinion, would impair the subject's ability to respond to vaccination.
* Severe hypersensitivity to any vaccine (anaphylaxis, angioedema, bronchospasm, or laryngospasm).
* History of asthma, chronic obstructive pulmonary disease, or other current/residual disease of the lungs.
* Clinically significant abnormal laboratory tests.
* Current smoker.
* Any known allergies to sodium succinate, Tween-20 (a detergent), aluminum hydroxide, or kanamycin.
* Previously received ricin toxin vaccine or has antibodies to ricin toxin proteins.
* Receipt of licensed vaccines within 30 days prior to the start of the study or plans to receive other vaccines during the initial 9 months of the study (the only exceptions are the inactivated influenza vaccine that can be received at least 30 days after RVEc Dose 3).
* Receipt of investigational drug/test product within 30 days prior to entry or within the initial 9 months of the study.
* Females: Pregnant or breastfeeding.
* Enrolled in another greater than minimal risk study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip R Pittman, MD, MPH, Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- Department of Clinical Research, U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

REFERENCES:
- [Result] Pittman PR, Reisler RB, Lindsey CY, Guerena F, Rivard R, Clizbe DP, Chambers M, Norris S, Smith LA. Safety and immunogenicity of ricin vaccine, RVEc, in a Phase 1 clinical trial. Vaccine. 2015 Dec 16;33(51):7299-7306. doi: 10.1016/j.vaccine.2015.10.094. Epub 2015 Nov 3. PMID 26546259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 10 | 10 | 10
Completed | 10 | 10 | 10 (The original trial design was modified to limit the number of vaccinations in Group 3 to 1 dose.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (8.19) | 35.0 (7.62) | 32.2 (8.13) | 34.3 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 7 | 6 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 9 | 10 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 10 | 9 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccinated Subjects Any Averse Events and by Location and Severity
Time Frame: Days 1, 3, 7, 14, and 28 after each vaccination and at 6 and 9 months
Population: Safety population: any subject receiving a vaccination
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 10 | 10
participants
  Any adverse events | 10 | 10 | 9
  Local life-threatening | 0 | 0 | 0
  Local severe | 1 | 0 | 0
  Local moderate | 1 | 0 | 0
  Local mild | 7 | 8 | 2
  Systemic life-threatening | 0 | 0 | 2
  Systemic severe | 3 | 2 | 2
  Systemic moderate | 7 | 8 | 5
  Systemic mild | 10 | 10 | 8

2. Secondary Outcome: Over Response Rates and Comparisons for ELISA and TNA Titers
Description: Overall response is defined as a subject having a response at any time after vaccination. A response is defined as subjects who developed total ELISA IgG titers (≥ 1:500) and TNA anti-ricin toxin-neutralizing antibody titers (≥ 1:50) at each scheduled time point for which blood samples were taken for each group and over the entire study period to study completion.
Time Frame: Day 7, 14, 28, 35, 42, 56, 63, 70, 84, month 6, 9, and 12
Population: Per-protocol population. Only observations or specimens collected according to the protocol were included in the immunogenicity analyses.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 10 | 10 | 10
participants
  ELISA | 10 | 6 | 6
  TNA | 5 | 0 | 1

ADVERSE EVENTS:
Time Frame: 9 months
Description: Safety population: any subject receiving a vaccination
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=10) | Group 2 (N=10) | Group 3 (N=10)
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 3 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Injection site pain (General disorders) | 7 | 8 | 1
Cyst (General disorders) | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0
Injection site papule (General disorders) | 1 | 0 | 0
Blood urea increased (Investigations) | 3 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (General disorders) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Investigations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 5 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0
Urine leukocyte esterase (Investigations) | 0 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 3
White blood cells urine (Investigations) | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood testosterone decreased (Investigations) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diastolic hypertension (Vascular disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes